CLINICAL TRIAL: NCT06012292
Title: Effect of Mobile Phone Addiction With Forward Head Posture on Pain and Cervical Functions
Acronym: FHP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amal Mohammed Bahgat Fayed, principle investigator Amal mohammed bahgat fayed, Cairo University
Other Study IDs: P.T.REC/012/004269
Record Dates: First submitted 2023-08-19; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-07

CONDITIONS: Forward Head Posture
Keywords: Cervical function, Forward head posture, Mobile phone addiction, Pain
MeSH Terms: conditions — Technology Addiction; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A Not addicted to mobile phone: Addicted to mobile phone less than four hours per day.
- Group B addicted to mobile phone: Addicted to mobile phone more than four hours per day.

SUMMARY:
to investigate the effect of mobile phone addiction with forward head posture on the endurance of deep neck flexor muscles, respiratory functions, pain pressure threshold , and neck functional disability level.

DETAILED DESCRIPTION:
Nowadays, the mobile phone has become an important requirement. The number of mobile phone users and the duration of mobile phone use are increasing rapidly, and the side effects can be detrimental one of them is forward head posture.

Prolonged use of the mobile phone has also affected posture, resulting in many musculoskeletal disorders or improper posture. Neck posture, particularly in a sitting position, is regarded an essential contributing factor to the development and long-term maintenance of cervical pain and headache. Neck flexed posture increased due to the frequent use of the relatively small screen of a mobile phone compared to that of a desktop computer. Constant use may also have unexpected consequences: increased stress on the cervical spine.

Forward head posture (FHP) is the most common side effect of prolonged, sustained mobile and tablet use. This leads to extension at atlantooccipital (C1 to C2) joints with flexion of lower cervical spine (C4 to C7) and flattening of mid cervical lordosis which cause joint dysfunction associated with negative affection of lung function, abnormal afferent information affecting the tonic neck reflex and encourages the gradual adaptation of FHP.

ELIGIBILITY:
Inclusion Criteria:

1. Forward head with craniovertebral angle less than 50 degree.
2. Both sexes will participate in this study.
3. Their age will be ranging from 18-40years (Molaeifar et al., 2021).
4. Body mass index is ranged from 18-25 kg /m2 (Molaeifar et al., 2021).
5. Area of mobile phone is 17 × 8cm.
6. Participants will be randomly allocated into 2 groups, group (A) should not have addicted to mobile phone and group (B) should have addicted to mobile phone.

Exclusion Criteria:

1. Previous cervical operation.
2. Musculoskeletal disorders such as cervical spine fracture, myelopathy, spinal cord tumor.
3. Neurological conditions that affected head, neck, and upper limbs.
4. Cervical disc or spondylosis.
5. Respiratory diseases such as Restrictions in lung function.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult both gender males and females, normal BMI, normal and forward head posture participants, addicted and not addicted to mobile phoine will be included in the study.
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold | one week
  Pain pressure threshold will be measured by pressure algometer
Respiratory functions | one week
  Respiratory functions including tidal volume and total lung capacity will be measured by incentive spirometer

SECONDARY OUTCOMES:
Endurance of deep neck flexor muscles | one week
  Endurance of deep neck flexor muscles will be measured by pressure biofeedback unit stabilizer
Neck functional disability level | one week
  Neck functional disability level will be measure by Copenhagen Neck Functional Disability scale Arabic version

CONTACTS AND LOCATIONS:
Locations (1):
- Amal Mohammed Bahgat Fayed, Beheira, Egypt